CLINICAL TRIAL: NCT06709729
Title: Switch of Open-source Automated Insulin Delivery System - AndroidAPS to Commercially Available AID Systems in Type 1 Diabetes: the Extension of the CODIAC Study
Brief Title: Switch of AndroidAPS to Commercially Available AID Systems
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: General University Hospital, Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CODIAC Extension
Record Dates: First submitted 2024-11-02; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Insulin Pump; Closed-loop hybrid system; Continuous Glucose Monitoring; Automated Insulin Delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Control-IQ or Smartguard system (Experimental): Patients with use of the Control-IQ system or Smartguard system (closed-loop hybrid system) and previous users of AndroidAPS (closed-loop hybrid system)
  Interventions: Device: Insulin pump with closed-loop system

INTERVENTIONS:
Device: Insulin pump with closed-loop system — Device: Usage of Insulin pump t:slim X2 with Control-IQ technology or MiniMed 780G with Smartguard technology in previous users of AndroidAPS
  Other Names: Insulin pump t:slim X2 with Control-IQ technology; Insulin pump MiniMed 780G with Smartguard technology in previous users of AndroidAPS

SUMMARY:
The aim of the study was to investigate the switch between open-source automated insulin delivery system (OS-AID) - AndroidAPS (AAPS) and commercially available AID systems - Control-IQ (CIQ) and MiniMed 780G (780G) in extended follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes diagnosed >2 years
* ≥ 18 years old
* written informed consent prior to starting study related activity
* previous user of AndroidAPS at least for 3 months

Exclusion Criteria:

* nonadherence to the current treatment regimen
* lactation
* pregnancy
* intending to become pregnant during study
* concomitant therapy influencing glucose metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of time in target ranges | 14 weeks
  3.9-10.0 mmol/L [70-180 mg/dL]

SECONDARY OUTCOMES:
Percentage of time in hypoglycemic range | 14 weeks
  <3.9 mmol/L [70 mg/dL] and <3.0 mmol/L [54 mg/dL]
Percentage of time in hyperglycemic range | 14 weeks
  >10,0 mmol/L [180 mg/dL] and >13,9 mmol/L [250 mg/dL]
Percentage of time in tight range | 14 weeks
  3.9 mmol/L-7.8 mmol/l [70 mg/dL - 140 mg/dL]
Changes in glycemic variability | 14 weeks
  Expressed as the coefficient of variation
Icidence of severe hypoglycaemia | 14 weeks
  Requiring third-party assistance to treat
Changes in glycated haemoglobin (HbA1c) | 14 weeks
  Differences between HbA1c values in the initial period and after follow-up
Hypoglycemia Attitudes and Behavior Scale (HABS) | 14 weeks
  This validated questionnaire contains in total 14 questions that highlights two critical dimensions of hypoglycemia related concerns (anxiety and avoidance) and one positive dimension (confidence). 14 items use Likert scales from 1 to 5, total score from 14 to 70, the higher total score means worse outcome.
Diabetec distress as assessed by validated questionnaire | 14 weeks
  The DDS17 yields a total diabetes distress score plus 4 subscale scores, each addressing a different kind of distress - Emotional Burden, Physician Distress, Regimen Distress, Interpersonal Distress. Scores in total and each subscales range between 1-21, higher scores denote higher distress.
The 5-item World Health Organization well-being index as assessed by validated questionnaire | 14 weeks
  This questionnaire contains in total 5 questions. Scores in total range between 0-25, higher scores denote higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Soupal, Principal Investigator — 3rd Department of Internal Medicine, 1st Faculty of Medicine, Charles University
Locations (1):
- 3rd Department of Internal Medicine, 1st Faculty of Medicine, Charles University, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hajos TR, Pouwer F, Skovlund SE, Den Oudsten BL, Geelhoed-Duijvestijn PH, Tack CJ, Snoek FJ. Psychometric and screening properties of the WHO-5 well-being index in adult outpatients with Type 1 or Type 2 diabetes mellitus. Diabet Med. 2013 Feb;30(2):e63-9. doi: 10.1111/dme.12040. PMID 23072401
- [Background] Do QD, Haskova A, Radovnicka L, Konecna J, Horova E, Parkin CG, Grunberger G, Prazny M, Soupal J. Comparison of Control-IQ and open-source AndroidAPS automated insulin delivery systems in adults with type 1 diabetes: The CODIAC study. Diabetes Obes Metab. 2024 Jan;26(1):78-84. doi: 10.1111/dom.15289. Epub 2023 Sep 25. PMID 37743832
- [Background] Haskova A, Radovnicka L, Petruzelkova L, Parkin CG, Grunberger G, Horova E, Navratilova V, Kade O, Matoulek M, Prazny M, Soupal J. Real-time CGM Is Superior to Flash Glucose Monitoring for Glucose Control in Type 1 Diabetes: The CORRIDA Randomized Controlled Trial. Diabetes Care. 2020 Nov;43(11):2744-2750. doi: 10.2337/dc20-0112. Epub 2020 Aug 28. PMID 32859607
- [Background] Soupal J, Petruzelkova L, Flekac M, Pelcl T, Matoulek M, Dankova M, Skrha J, Svacina S, Prazny M. Comparison of Different Treatment Modalities for Type 1 Diabetes, Including Sensor-Augmented Insulin Regimens, in 52 Weeks of Follow-Up: A COMISAIR Study. Diabetes Technol Ther. 2016 Sep;18(9):532-8. doi: 10.1089/dia.2016.0171. Epub 2016 Aug 2. PMID 27482825
- [Background] Soupal J, Petruzelkova L, Grunberger G, Haskova A, Flekac M, Matoulek M, Mikes O, Pelcl T, Skrha J Jr, Horova E, Skrha J, Parkin CG, Svacina S, Prazny M. Glycemic Outcomes in Adults With T1D Are Impacted More by Continuous Glucose Monitoring Than by Insulin Delivery Method: 3 Years of Follow-Up From the COMISAIR Study. Diabetes Care. 2020 Jan;43(1):37-43. doi: 10.2337/dc19-0888. Epub 2019 Sep 17. PMID 31530663